CLINICAL TRIAL: NCT05776862
Title: A Pilot Study Testing Benefits of Ursolic Acid (UA) as a Countermeasure To Myopenia and Insulin Resistance in Chronic Spinal Cord Injury (SCI)
Brief Title: Study Testing Benefits of Ursolic Acid (UA) as a Countermeasure To Myopenia and Insulin Resistance in Chronic Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20221142; COPBC (Other: State of Florida)
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Tetraplegia; Paraplegia; Muscle Loss; Atrophy, Muscular; Insulin Resistance
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia; Muscular Atrophy; Insulin Resistance | interventions — Ursolic Acid; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UA and exercise in paraplegia group (Experimental): Participants will take UA 4 capsules twice daily for 12 weeks while participating in an exercise program, 3 times per week.
  Interventions: Drug: Ursolic Acid; Other: Strength Training
- UA in tetraplegia group (Experimental): Participants will take UA 4 capsules twice daily for 12 weeks
  Interventions: Drug: Ursolic Acid

INTERVENTIONS:
Drug: Ursolic Acid — Subjects will take an oral 400mg (8 capsules - 4 in the morning/200mg and 4 at night/200mg) supplement of UA every day for 12 weeks.
Other: Strength Training — Subjects will perform 3 sets of 10 repetitions of concentric and eccentric upper body exercises (bicep curls and tricep extensions) each session. Each session will last approximately 10-15 minutes of weightlifting with a 2-minute rest period between sets. The arm selected for exercise will be randomized.
  Arms: UA and exercise in paraplegia group

SUMMARY:
This study will evaluate if Ursolic Acid supplementation may be effective in reducing muscle loss and improving blood sugar control in the SCI community.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals with paraplegia having chronic (> 1 year) motor-complete and incomplete (AIS A/B/C) injuries from T2-T8
2. Male and female individuals wi4.th chronic (> 1 year) motor-complete and incomplete (AIS A/B/C) injuries from C4-C7

Exclusion Criteria:

1. Pregnant or planning to become pregnant
2. Women who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami - Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UA and Exercise in Paraplegia Group | UA in Tetraplegia Group
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UA and Exercise in Paraplegia Group | UA in Tetraplegia Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (14.8) | 37.8 (9.1) | 37.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Mass Using Dual X-ray Absorptiometry (DXA)
Description: Changes in muscle mass in grams as measured by Dual X-ray Absorptiometry
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | UA and Exercise in Paraplegia Group | UA in Tetraplegia Group
Number analyzed (Participants) | 4 | 4
grams | -183.00 (2642.65) | 1434.00 (1885.21)

2. Primary Outcome: Changes in Peak Isokinetic Strength
Description: Peak strength (peak torque in ft-lb) of both arms at 90 degrees range of motion will be tested in elbow flexion and extension (at 60 deg/s) on a Biodex dynamometer
Time Frame: Baseline, 12 weeks
Population: Only paraplegia group participated in this outcome measure, per protocol.
Measure: Mean (Standard Deviation); unit: ft-lb
Arm/Group | UA and Exercise in Paraplegia Group
Number analyzed (Participants) | 4
ft-lb
  Involved arm flexion | 5.58 (3.55)
  Uninvolved arm flexion | 1.83 (3.01)
  Involved arm extension | 3.05 (7.33)
  Uninvolved arm extension | 9.63 (3.00)

3. Primary Outcome: Changes in Fasting Insulin Resistance (IR)
Description: Changes in IR using Homeostatic Model of Assessment (HOMA) v2 model estimates steady state beta cell function and insulin sensitivity as percentages of a normal reference population. The change in resting IR will be measured by (fasting serum glucose*fasting serum insulin/22.5). Lower values indicate a higher degree of insulin sensitivity.
Time Frame: Baseline, 12 weeks
Population: Only the tetraplegia group participated in this outcome measure, per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UA in Tetraplegia Group
Number analyzed (Participants) | 4
score on a scale | 1.6125 (2.70)

4. Primary Outcome: Changes in Glucose Disposal
Description: Changes in glucose disposal will be measured by the Oral Glucose Tolerance Test (OGTT) using Trutol glucose solution of 75 grams. The rates of glucose disposal will be defined by the area under the glucose challenge curve (AUC).
Time Frame: Baseline, 12 weeks
Population: Only the tetraplegia group participated in this outcome measure, per protocol
Measure: Mean (Standard Deviation); unit: AUC (mg-dL/120 minutes)
Arm/Group | UA in Tetraplegia Group
Number analyzed (Participants) | 4
AUC (mg-dL/120 minutes) | 930.75 (2327.13)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | UA and Exercise in Paraplegia Group | UA in Tetraplegia Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UA and Exercise in Paraplegia Group (N=5) | UA in Tetraplegia Group (N=5)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UA and Exercise in Paraplegia Group (N=5) | UA in Tetraplegia Group (N=5)
changes in urine (Renal and urinary disorders) | 0 (0) | 1 (1) — change in urine color, smell, consistency
increased gas or bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT05776862/Prot_SAP_000.pdf